CLINICAL TRIAL: NCT00463463
Title: Phase III Stidy of Zevalin And BEAM Compared With BEAM Alone Prior to Autologous Hematopoietic Steem Cell Transpl. in Pts Relapse of Non-Hodgkins Lymphoma
Brief Title: Zevalin and BEAM High-dose Chemotherapy Compared With BEAM Alone as Conditioning Regimen in Patients With Chemosensitive Relapse of Non-Hodgkin's Lymphoma
Acronym: Zevalin
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sor451107ctil
Record Dates: First submitted 2007-04-19; First posted 2007-04-20 (Estimated); Last update posted 2012-07-12 (Estimated); Status verified 2007-02

CONDITIONS: Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — ibritumomab tiuxetan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: 90Yttrium Ibritumomab Tiuxetan (Zevalin)

SUMMARY:
High-dose chemotherapy and autologous stem-cell transplantation have an established role in the treatment of aggressive Non-Hodgkin's lymphoma (NHL) when refractory to first line chemotherapy or after relapse. The PARMA study randomized 109 patients, with chemo-sensitive relapse and no marrow involvement to receive, following the initial salvage regimen, high-dose chemotherapy versus continuous standard dose chemotherapy. 5-year progression-free survival was 46% in the transplant group compared with 12% in the chemotherapy group. Results are significantly inferior in patients with multiply relapsed or chemo-refractory disease with only 0-20% of patients achieving long-term disease control with autologous transplantation. Thus a large proportion of patients with refractory and relapsing disease are not cured with currently available transplantation methods and newer approaches are required.

Rituximab is the first monoclonal antibody approved for clinical use. It is an anti CD20 antibody with high response rate in the treatment of follicular lymphoma and increases response rate in aggressive lymphoma when combined with chemotherapy. It is well tolerated with minimal side effects. However tumors may escape rituximab sensitivity by loss of antigen, poor access of antibody to bulky or poorly vascularized tumors, or failure of host effectors to eliminate antibody binding tumor cells. Lymphoma cells are inherently and exquisitely sensitive to radiation. Radioimmunotherapy uses monoclonal antibodies conjugated with a radioactive isotope to target radiation directly to tumor cells. Ibritumomab is the parent murine anti CD20 antibody witch targets the same epitope as rituximab. Tiuxetan is a chelator covalently linked to the antibody which chelates the isotope 90Yttrium to form the active radioconjugate Zevalin. 90Yttrium is a pure high-energy beta emitter with a relatively short half time (64 hours) and a path length of 5 mm. These properties make it an ideal isotope for radioimmmunotherapy. The high energy and long beta path are advantageous in treating bulky, poorly vascularized tumors, and tumors with heterogeneous antigen expression as neighboring tumor cells can be hit by cross fire from tumors binding the radioconjugate. Pure beta emission limits radiation to the patient body and is safe for the surrounding allowing simple outpatient care, no need for patient isolation or shielding. Biodistribution is predictable, eliminating the need for dosimetry. Initial studies showed that Zevalin has a favorable toxicity profile and is more effective than rituximab in patients with follicular and transformed non-Hodgkin's lymphoma, and studies are currently performed in aggressive lymphoma.

There are initial phase I-II studies combining radioimmunotherapy with high-dose chemotherapy and autologous stem-cell transplantation with promising results. We conducted a phase II study of fixed-dose Zevalin at 0.4 mCi/kg with BEAM high-dose chemotherapy in patients with chemo-refractory disease. So far, 23 patients were included. With a median follow-up of 17 months the estimated progression-free survival was 52% compared with 0-20% expected in patients with multiply relapsed and chemo-refractory disease. Based on these data and data from other groups we expect that the addition of Zevalin to standard high-dose chemotherapy will improve transplantation outcomes in patients with standard-risk chemosensitive disease, as well. This study will randomize patients to Zevalin-BEAM versus BEAM alone to determine the potential of Zevalin radioimmunotherapy to improve outcome of autologous stem-cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with CD20 positive aggressive non-Hodgkin's lymphoma, either diffuse large B-cell or transformed follicular lymphoma as confirmed by a pathological biopsy report.
2. Patients who are candidates for stem-cell transplantation due to refractory disease to first line chemotherapy or relapsing disease and comply with standard transplant eligibility criteria.
3. Patients must have chemo-sensitive disease achieving at least partial response to salvage chemotherapy.
4. Patients were given up to 2 lines of therapy, initial treatment and one salvage treatment. Local radiation therapy for consolidation is not considered a line of therapy.
5. Age less than physiologic 65 years.
6. Patients with an adequate autologous stem cell collection for transplantation (>2.5 x 106 CD34+ cells/kg). Backup collection is preferable but not obligatory.
7. Patients must sign written informed consent.
8. Adequate birth control in fertile patients.
9. All prior chemotherapy completed at least three weeks before study treatment

Exclusion Criteria:

1. Chemo-refractory disease or more than 2 prior therapies
2. Bilirubin > 3.0 mg/dl, transaminases > 3 times upper normal limit
3. Creatinine > 2.0 mg/dl
4. ECOG-Performance status < 2
5. Uncontrolled infection
6. Pregnancy or lactation
7. Abnormal lung diffusion capacity (DLCO < 40% predicted)
8. Severe cardiovascular disease
9. Chemo-refractory disease as determined by less than partial response to salvage chemotherapy.
10. active CNS disease involvement
11. Pleural effusion or ascites > 1 liter
12. Known hypersensitivity to rituximab
13. Psychiatric conditions/disease that impair the ability to give informed consent or to adequately co-operate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2007-04

CONTACTS AND LOCATIONS:
Overall Officials: Arnon Nagler, MD, Principal Investigator — Division of Hematology and Bone Marrow Transplantation
Locations (1):
- Soroka Universuty Medical Center, Beersheba, Israel